CLINICAL TRIAL: NCT07358611
Title: ELectrocardiographic Imaging-guided Substrate Ablation in Patients With Atrial Fibrillation - a PILOT Study of a Personalized Therapy
Brief Title: Non-invasive Mapping-Guided Atrial Fibrillation Ablation
Acronym: ELISA-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2024/1096
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial fibrillation; Catheter ablation; Atrial fibrillation drivers; Personalized atrial fibrillation therapy; Electroanatomical mapping; Electrocardiographic imaging; Body surface mapping
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-invasive mapping-guided ablation (Experimental): In this arm patients undergo a personalized ablation approach: In addition to conventional pulmonary vein isolation, additional target regions will be ablated based on non-invasive global mapping.
  Interventions: Procedure: Non-invasive mapping-guided ablation

INTERVENTIONS:
Procedure: Non-invasive mapping-guided ablation — The study intervention consists of
  1. Empirical pulmonary vein isolation (current standard of care) plus
  2. A personalized ablation approach targeting up to three additional atrial regions which harbour critical AF-perpetuating sources:
     * Target regions are selected based on the spatiotemporal Stability of Atrial High-Rate Activity (SAHRA) using a non-invasive global mapping system (Acorys, Corify Care).
     * Selected target regions displaying stable high-rate activity are isolated or homogenized according to predefined regional borders based on the 15-segment bi-atrial model of the EHRA and EACVI Clinical Consensus on Standardized Atrial Regionalization (Althoff et al. 2025).

SUMMARY:
The goal of this pilot study is to test if noninvasive global mapping can guide catheter ablation defining personalized targets and improve the therapy of atrial fibrillation. It will also test the safety of such an approach. The main questions it aims to answer are:

* Does ablation of targets defined by noninvasive global mapping improve rates of acute atrial fibrillation termination?
* Does such a personalized ablation approach reduce arrhythmia recurrence rates? Researchers will compare the results of the personalized ablation approach with comparable patients that had undergone a conventional "empirical" ablation approach (pulmonary vein isolation).

Participants will:

* Undergo a personalized catheter ablation approach employing both a noninvasive global mapping system and a conventional intracardiac mapping system
* Visit the clinic 3, 6 and 12 months after ablation for clinical follow-up
* Schedule a telephone visit 9 and 24 months after ablation for clinical follow-up

DETAILED DESCRIPTION:
The aim of this study is to test the feasibility and potential of a personalized, non-invasive mapping-guided ablation approach in patients with persistent atrial fibrillation (AF), who are unlikely to benefit from empirical pulmonary vein isolation alone. As a pilot study, it is designed to assess feasibility and procedural efficacy and potential signals of harm.

General Strategy:

Patients with persistent AF planned for catheter ablation are eligible in case of left atrial enlargement.

The study intervention consists of

1. Empirical pulmonary vein isolation in all patients (current standard of care).
2. A personalized ablation approach targeting up to three additional atrial regions which harbour critical AF-perpetuating sources:

   * Target regions are selected based on the spatiotemporal Stability of Atrial High-Rate Activity (SAHRA) using a non-invasive global mapping system (Acorys, Corify Care).
   * Selected target regions displaying stable high-rate activity are isolated or homogenized according to predefined regional borders based on the 15-segment bi-atrial model of the EHRA and EACVI Clinical Consensus on Standardized Atrial Regionalization (Althoff et al. 2025).

ELIGIBILITY:
Inclusion Criteria:

Ablation-naïve patients with:

1. Persistent AF planned for catheter ablation plus
2. Left atrial enlargement (LA diameter ≥45 mm or LA volume index ≥35ml/m2 or LA area ≥20 cm2)

Exclusion Criteria:

* Previous cardiac ablation
* Age <18 years
* Pregnancy or lactation
* Previous stroke/TIA
* Severe left ventricular dysfunction (LVEF <35%)
* Renal failure (GFR <30 ml/min)
* Dermal disease or hypersensitivity predisposing for skin irritation or exanthema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute AF termination | Procedural
  Rate of acute AF termination (ro sinus rhythm or conversion into an organized atrial tachycardia) upon ablation

SECONDARY OUTCOMES:
Proportion of patients with arrhythmia-free survival | Days 91 to 365 post-ablation
  Absence of any atrial tachyarrhythmia (atrial fibrillation [AF], atrial flutter [AFL] or atrial tachycardia [AT]) between days 91 and 365 post ablation. AF, AFL or AT will qualify as a recurrence after ablation if it lasts 30 s or longer.
Proportion of patients with AF-free survival | Days 91 to 365 post-ablation
  Absence of atrial fibrillation [AF] between days 91 and 365 post ablation. AF will qualify as a recurrence after ablation if it lasts 30 s or longer
Rate of procedure-related complications | Day 0 to 30 post-ablation
  Composite safety endpoint composed of:
  * cardiac tamponade requiring drainage
  * persistent phrenic nerve palsy lasting >24 hours
  * serious vascular complications requiring intervention
  * stroke/TIA
  * atrioesophageal fistula
  * death

CONTACTS AND LOCATIONS:
Overall Officials: Till F Althoff, M.D., Principal Investigator — German Heart Center of the Charite, Berlin; Ivo Roca-Luque, M.D., Ph.D., Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, University of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Data underlying published results will be provided upon reasonable request

REFERENCES:
- [Background] Invers-Rubio E, Hernandez-Romero I, Reventos-Presmanes J, Ferro E, Guichard JB, Regany-Closa M, Pellicer-Sendra B, Borras R, Prat-Gonzalez S, Tolosana JM, Porta-Sanchez A, Arbelo E, Guasch E, Sitges M, Brugada J, Guillem MS, Roca-Luque I, Climent AM, Mont L, Althoff TF. Regional conduction velocities determined by noninvasive mapping are associated with arrhythmia-free survival after atrial fibrillation ablation. Heart Rhythm. 2024 Sep;21(9):1570-1580. doi: 10.1016/j.hrthm.2024.04.063. Epub 2024 Apr 16. PMID 38636930